CLINICAL TRIAL: NCT05803655
Title: Does Time From Ovulation Trigger To Oocyte Pick-Up Affect Intracytoplasmic Sperm Injection Outcomes? A Multi-Center Single-Blinded Randomized Controlled Trial Comparing 36 and 38 Hour Intervals
Brief Title: Outcomes of 36 vs 38 Hour Intervals From Ovulation Trigger To Oocyte Pick-Up:A Multi-Center Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Collaborators: Turkish Society of Reproductive Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021.267.IRB1.093
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-04

CONDITIONS: Infertility; IVF
Keywords: oocyte pick-up; in vitro fertilization; oocyte maturation; ovulation trigger; intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: The patient will be randomized to either ''36 hour'' or ''38 hour'' group on the day of ovulation trigger. According to her allocation, she will apply the injection. Except for the difference in the interval between ovulation trigger and oocyte pick-up procedure, women in both arms will undergo exactly the same treatment steps.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the head-nurse and the patient will not be masked, since one will randomize the patient to a group and give her instructions on how to use the medication, and the other will apply the injection herself.
  However, allocation will be concealed from the the laboratory team, treating physicians, outcome assessors and investigators. They will not be given information about when the patient applied the injection, and the patient will be instructed not to reveal information regarding her use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 36-Hour Group (Active Comparator): The women randomized to this group will undergo oocyte pick-up procedure 36 hours after the injection of the ovulation triggering agent.
  The choice for ovulation trigger agent is at the discretion of the treating physician. The intervention is not the drug but the interval.
  Interventions: Other: 36-hour duration between ovulation triggering and oocyte pick-up procedure
- 38-Hour Group (Experimental): The women randomized to this group will undergo oocyte pick-up procedure 38 hours after the injection of the ovulation triggering agent.
  The choice for ovulation trigger agent is at the discretion of the treating physician. The intervention is not the drug but the interval.
  Interventions: Other: 38-hour duration between ovulation triggering and oocyte pick-up procedure

INTERVENTIONS:
Other: 36-hour duration between ovulation triggering and oocyte pick-up procedure — 36-hour duration between ovulation triggering and oocyte pick-up procedure
  Arms: 36-Hour Group
Other: 38-hour duration between ovulation triggering and oocyte pick-up procedure — 38-hour duration between ovulation triggering and oocyte pick-up procedure
  Arms: 38-Hour Group

SUMMARY:
Women who undergo assisted reproduction technology (ART) treatment will be eligible for this study. The goal of this randomized clinical trial is to compare the outcomes of ART treatment between women who have 36 and 38 hours interval between the administration of ovulation trigger (ovulation trigger medication initiates oocyte maturation and makes it possible for the egg to be collected by aspiration, during a procedure called oocyte pick-up, OPU) and OPU. The main questions it aims to answer are, does prolonging the trigger-OPU interval to 38-hours improve:

1. Primarily:

   •Ratio of metaphase-2 oocytes to total number of follicles
2. Secondarily:

   * Maturation rate
   * Fertilization rate
   * Blastulation rate
   * Premature ovulation rate
   * Positive pregnancy test rate
   * Clinical pregnancy rate
   * Live birth rate

compared to 36-hours interval?

DETAILED DESCRIPTION:
1.0 STUDY POPULATION AND PATIENT SELECTION Women undergoing ART treatment at the participating centers will be invited to enroll in the study. Each patient will be able to participate only once with a single oocyte pick-up (OPU) cycle and embryos obtained from this cycle. Details of inclusion and exclusion criteria are described in the ''Eligibility'' section.

2.0 RANDOMIZATION METHOD AND ALLOCATION CONCEALMENT Couples who meet the study criteria will be informed about the study when they start treatment and will be given time to decide. On the day of ovulation trigger administration, patients who give written informed consent will be enrolled and randomized to one of the study groups (36 or 38 hours) by the nurse-in-charge. The patient will be instructed about the administration time by the nurse. Randomization information will not be shared with clinicians, laboratory team or other employees in the clinic throughout the study. The patient will also be asked not to share this information with anyone from the staff.

Randomization will be performed online in real time by a professional third-party company whose services meet international regulatory guidelines. The randomization sequence will be stratified by treatment center, female age group (18-27, 28-34, 35-37, 38-40, 41-42), anticipated embryo transfer day (day 3 and day 5), and plan to utilize preimplantation genetic testing for the embryos. Randomized blocks of varying size (4,6, or 8) will be created to ensure a similar number of patients among the study groups in each stratum during and at the end of the study.

3.0. TREATMENT PROTOCOLS The intervention in this study is the time between the ovulation trigger and the OPU procedure. Therefore, each clinic will apply their own routine treatments and make their own choices regarding the protocols/drugs/materials and/or procedures to be used.

3.1. Controlled Ovarian Hyperstimulation(COH) and Triggering of Oocyte maturation One of three protocols for COH can be applied according to the preference of the clinician: Antagonist protocol, progestin-primed ovarian stimulation, or agonist protocol.

Once the decision to trigger oocyte maturation is made, the nurse-in-charge will randomize the patient.

3.2. Oocyte collection(OPU) procedure On the day of OPU, the nurse-in-charge will confirm and note the time the patient administered the medication. She will then record the OPU start time and assess adherence to the protocol. The time of OPU will be based on the hour and minute when the first follicle was aspirated and recorded.

The total number of follicles larger than 10 mm on ultrasonography performed before OPU and the presence of premature ovulation signs will be recorded. The needle and solution routinely used by the clinic will be used for OPU. All follicles >10 millimeters in diameter will be aspirated.

3.3. Fertilization, Embryo Culture and Embryo Transfer All mature oocytes obtained by OPU will be fertilized by intracytoplasmic sperm injection (ICSI). After fertilization, oocytes/embryos will be cultured according to the standard protocols of the center.

Embryo(s) will be transferred fresh or frozen-thawed at the clinician's discretion. Preparation for frozen-thawed embryo transfers will be performed as a natural, modified natural, or artificial cycle, again at the clinician's discretion.

Embryo transfers will be performed under ultrasonography guidance at the cleavage or blastocyst stage(day 3 or day 5) according to the clinician's preference and clinic protocol. One or two embryos will be transferred in accordance with the Ministry of Health regulations. Luteal phase support will be provided in accordance with the routine treatment of each clinic.

4. EVALUATION OF RESULTS Primary and secondary outcome measures are described in the ''Outcome Measures'' section.

5. DATA COLLECTION AND MANAGEMENT 5.1. Data Collection Study data will be entered daily into the electronic data collection (EDC) form of the study. EDC forms are filled online in real time and stored by a professional third-party company whose services will meet compliance certifications worldwide such as U.S. Food and Drug Administration (FDA) Code of Federal Regulations (CFR) Part 11; The General Data Protection Regulation(GDPR) European Union(EU); International Conference on Harmonisation Good Clinical Practice (ICH GCP); The Health Insurance Portability and Accountability Act, United States(HIPAA, US); the International Organization for Standardization(ISO) 27001; ISO 9001, and will align with Good Clinical Practice(GCP); Health Level 7,Fast Health Interoperability Resources(HL7 FHIR) and other regulatory guidelines.

Each quarter, a member of the study team will compare the consistency between the data entered in the clinic records and the EDC form. Preferably and if feasible, all actual files in the center and the EDC form will be compared; if this is not feasible, a part of the files (at least 50%) will be randomly selected and compared.

5.2. Data Collection Period The results will be evaluated after the information of the last included patient has been completed. At this point, all entries into the database will be confirmed as complete and only then will the randomization code be broken and the data analysis process will begin.

5.3. Electronic database, data entry and quality control An electronic database will be established to record the study data. This database will be maintained by an external organization capable of meeting the security, confidentiality, backup and quality standards to be defined. Study data will be entered daily into the study EDC form by authorized study coordinators and the database will be updated and backed up in real time. Only authorized persons will have access to the database, and each person will be authorized to see, see/write, or see/write/modify data according to their role. Data modification or deletion will require the approval of at least two authorized persons, and these changes will be tracked and justified.

Quality control will be performed quarterly during the study period. In each period, the original patient follow-up files of preferably all(or if this is not feasible, randomly selected one-half) of the participants accumulated at each center will be compared with the data in the database. The acceptable error rate is zero for the primary outcome measure and less than 5% for other variables. In any control, when the discrepancy between the original forms and the database in a center exceeds 5%, the original records of that center will be compared with all entries of that center in the database and data cleaning will be performed. In order to minimize data entry errors and omissions, mandatory fields to be filled in the electronic data collection form will be determined and the form will not be saved to the system without filling in these fields; similarly, the software will not allow entering a value other than the expected values for each parameter.

6. STATISTICAL EVALUATION 6.1. Sample Size Calculation Considering that the rate of metaphase-2 oocytes obtained per aspirated follicle during OPU in our clinic is 57%, calculations based on the hypothesis that an absolute 10% increase in this rate will be achieved with the intervention to be tried, it was revealed that a total of 770 patients should be randomized at 80% power and 5% alpha error level. Assuming that approximately 10% of patients would drop out of the study during follow-up, 850 patients would be randomized. Six centers will participate in the study and it is thought that this number will be reached in 1 year with the anticipated study tempo.

In the first two interim analyses, this sample size can be revised according to the efficacy data obtained in the study so far, provided that the same alpha error and statistical power rates are maintained.

6.2. Handling of Missing Data Patients with missing data will not be excluded from the analyses, but will be included in the intention-to-treat analysis. When there are patients with missing outcome measure data, sensitivity analysis will be performed to calculate how the results may change under different scenarios.

6.3. Statistical Analysis Plan Results will be evaluated primarily according to the intention-to-treat principle. Dropping out of follow-up will not mean dropping out of the study. The time between the time of administration of the drug used for oocyte maturation and OPU will be recorded as not occurring in accordance with the group to which the patient was randomized. Thirty minutes before and after the target (36 hours ± 30 minutes or 38 hours ± 30 minutes) will be considered to be within the protocol.

On the other hand, if for any reason, the time between drug administration-OPU does not comply with the protocol to which the patient was assigned according to the above criteria, the patient will not be excluded from the study; the time in question will be recorded in hours and minutes and included in the per-protocol analysis to be performed according to this time. Per protocol analysis will be performed according to one-hour time intervals.

Comparisons of continuous variables between groups will be made by t-test or Mann-Whitney U test according to the distribution characteristics of each variable, and comparisons of categorical variables will be made by chi-square and its derivatives.

The values of continuous variables in groups will be summarized with appropriate measures of central aggregation and dispersion, while the values of categorical variables will be expressed in absolute values and percentages.

Multivariable regression analysis will be performed for the effect of trigger-OPU time, female age, number of metaphase-2 oocytes microinjected, total number of embryos transferred on cumulative live birth.

6.3.1. Interim Analyses

Data for the primary and secondary outcome measures will be evaluated at 6-month intervals throughout the study period. The Peto-Haybittle stopping rule will be used in the interim analyses and a p < 0.01 for the primary outcome measure comparison will be required to stop the study early. The first interim analysis is planned to be performed when the first 80 patients are enrolled or 3 months later, whichever comes first.

7. SAFETY, ADVERSE EFFECTS AND RISKS Participants will be informed about the risks of the treatment and the expectation of success by providing an informed consent form for the study and an ART informed consent form.

The overall course of the study will be monitored at regular intervals by a Data and Safety Monitoring Board, including the rate of patient enrollment, compliance with the study protocol and the accumulated results. This safety board may recommend that the study be stopped early.

Study procedures are standard ART practice and no pharmaceutical agents or medical devices will be used outside of routine practice. Apart from the risks associated with ART itself, no additional medical risk or financial burden is expected to be associated with the study.

Serious adverse event(SAE) is defined as an event that causes death, threatens life, requires hospitalization or prolongs the duration of hospitalization, or causes permanent/significant incapacitation/disability. One of these is not expected to occur. A suspected unexpected serious adverse reaction(SUSAR) is defined as both an unexpected and serious adverse event. SAEs and SUSARs will be recorded and reported using SAE forms. If a SUSAR occurs, the form will be filled out immediately by the researcher and the Koç University Ethics Committee and the Data and Safety Monitoring Board will be informed immediately. The Ministry of Health will be informed within 7 days if the event is life-threatening and within 15 days if the event is not life-threatening.

ELIGIBILITY:
Inclusion Criteria:

* To undergo assisted reproductive technology (ART) treatment and planning to undergo embryo transfer procedure within 6 months of oocyte collection
* Female partner to be between 18-42 years old at the time of informed consent
* Both partners to consent to participate in the study and be legally eligible to give consent.

Exclusion Criteria:

* Female partner to have participated in the study previously.
* Female partner to have a body mass index of 35 kg/m2 or above.
* Female partner to have a systemic disease that may affect ART or pregnancy outcomes (e.g. antiphospholipid syndrome, severe liver dysfunction, diabetes mellitus, history of venous thrombosis, advanced renal or cardiac diseases).
* Presence of congenital uterine anomaly (1-Women whose uterine anomalies are surgically corrected are not excluded; 2- Arcuate uterus is not accepted as a congenital uterine anomaly).
* Presence of submucous or intramural fibroid that distorts the endometrial cavity.
* Diagnosis of stage 3 or 4 endometriosis in the female partner.
* Female partner planned to undergo double ovarian stimulation.
* Known karyotype anomaly in at least one of the partners.
* Diagnosis of azoospermia (no sperm cells in the ejaculate) in the male partner.
* History of recurrent implantation failure [defined according to the scoring system by Ata et al in 2021 available at https://bit.ly/3huVLOn (Ata B, Kalafat E, Somigliana E. A new definition of recurrent implantation failure on the basis of anticipated blastocyst aneuploidy rates across female age. Fertil Steril. 2021;116(5):1320-1327. doi:10.1016/j.fertnstert.2021.06.045].
* History of recurrent pregnancy loss [defined as a history of 2 or more biochemical/clinical pregnancy losses, in accordance with the European Society of Human Reproduction and Embryology(ESHRE) Guideline on the management of recurrent pregnancy loss issued on 1 February 2023, available at https://www.eshre.eu/Guidelines-and-Legal/Guidelines/Recurrent-pregnancy-loss.aspx].

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since ovarian stimulation, ovulation trigger and oocyte pick-up procedure can only be applied to females, we have to limit gender to female participants only.
Enrollment: 850 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ratio of metaphase-2 oocytes to total number of follicles | 1 day
  Number of metaphase-2 oocytes / total number of follicles >10mm prior to oocyte pick-up procedure

SECONDARY OUTCOMES:
Maturation rate | 2 days
  Metaphase-2 oocyte number / total number of oocytes
Fertilization rate | 2 days
  Number of two-pronuclei(2PN) embryos / number of metaphase 2 oocytes that underwent intracytoplasmic sperm injection
Cleavage rate | 4 days
  Number of cleavage stage embryos/number of 2PN embryos
Blastulation rate | 7 days
  Number of blastocyst stage embryos / number of 2PN embryos
Premature ovulation rate | 1 day
  Number of premature ovulation cases (Defined as detection of ovulation by ultrasound prior to oocyte pick-up procedure) / number of women enrolled
Positive Beta Human chorionic gonadotropin(Beta-hCG) test rate | 8 months
  Number of women with Positive serum Beta-hCG test (test will be performed 10 days after embryo transfer minimum) / total number of women enrolled
Clinical pregnancy rate | 8 months
  Number of women with clinical pregnancy (defined as intrauterine pregnancy with positive fetal heart beat in transvaginal ultrasound exam) / total number of women enrolled
Ongoing pregnancy rate | 8 months
  Number of women with pregnancy beyond 24th gestational week / total number of women enrolled
Live birth rate | 17 months
  Number of women who deliver at least one live fetus beyond 24th gestational week / total number of women enrolled
Miscarriage rate | 1 year
  Number of women negative fetal heart beat in transvaginal ultrasound exam before 24th gestational week / total number of women with clinical pregnancy
Biochemical pregnancy rate | 1 year
  Number of women with no sign of pregnancy during transvaginal ultrasound exam performed after a minimum of 30 days following embryo transfer / total number of women with positive Beta-hCG test
Ectopic pregnancy rate | 1 year
  Number of women with ectopic pregnancy / total number of women with positive Beta-hCG test

OTHER OUTCOMES:
Total oocyte number | 1 day
  Total number of oocytes after oocyte pick-up

CONTACTS AND LOCATIONS:
Overall Officials: Engin Turkgeldi, Assoc. Prof, Principal Investigator — Koç University; Baris Ata, Prof.Dr, Principal Investigator — Koç University
Locations (7):
- Turkey (Türkiye) (7):
  - Baskent University, Adana
  - Ankara University, Ankara
  - Hacettepe University, Ankara
  - Uludag University, Bursa
  - Koc University, Istanbul
  - Bahceci Fulya IVF Centre, Istanbul
  - VKF American Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available. However, upon reasonable request, anonymous data can be shared with interested parties.

REFERENCES:
- [Background] Ata B, Kalafat E, Somigliana E. A new definition of recurrent implantation failure on the basis of anticipated blastocyst aneuploidy rates across female age. Fertil Steril. 2021 Nov;116(5):1320-1327. doi: 10.1016/j.fertnstert.2021.06.045. Epub 2021 Jul 28. PMID 34332750
- See also: ESHRE Guideline on the management of recurrent pregnancy loss — https://www.eshre.eu/Guidelines-and-Legal/Guidelines/Recurrent-pregnancy-loss.aspx